CLINICAL TRIAL: NCT02898766
Title: Plasma Glucose and Insulin Response to Two Enteral Formulas in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response to Two Enteral Formulas in Persons With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16.17.CLI
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteral Nutrition Formula 1 (Active Comparator): Enteral Nutrition Formula
  Interventions: Other: Enteral Nutrition Formula
- Enteral Nutrition Formula 2 (Active Comparator): Enteral Nutrition Formula
  Interventions: Other: Enteral Nutrition Formula

INTERVENTIONS:
Other: Enteral Nutrition Formula

SUMMARY:
This will be a randomized, cross-over design. Subjects will be randomized to one of two interventions on two separate study days, 1 week apart.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 yrs
* Type 2 diabetes controlled with diet or diet and oral agent, with the exception of sulfonylureas such as glimepiride (Amaryl), glipizide, Glucotrol/GlucotrolXL) and glyburide (DiaBeta, Micronase, (Glynase Prestabs); meglitinides such as reaglinide (Prandin) and nateglinide (Starlix); and alphaglucosidase inhibitors such as acarbose (Precose) and miglitol (Glyset)
* Hemoglobin A1C less than 9.0%
* Fasting blood glucose less than 180 mg

Exclusion Criteria:

* Abnormal thyroid function
* Creatinine >2.0 mg/dL
* Potassium <3.5 mEq/L
* Gastrointestinal disease: ulcer, gastritis, diarrhea, gastroparesis, vomiting
* History of bypass surgery, midface trauma, esophageal varices, coagulation abnormalities
* Patients currently on any anti-coagulant medication
* Currently unstable diabetes or under treatment for cancer, heart disease, renal disease
* Unable to give informed consent or follow instructions
* Current insulin therapy or insulin therapy within the past month
* Patient who are pregnant
* Allergies to milk, fish oil or any component of the test product
* Patient who in the Investigators assessment cannot be expected to comply with treatment
* Currently participating or having participated in another clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose curve (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

SECONDARY OUTCOMES:
Area under the insulin curves (AUC 0-240) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
Insulinogenic index (Ins30/(Glu30)) | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes
AUC (0-30min) for insulin | Baseline, 10, 20, 30, 60, 90, 120, 150, 180, 210 and 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States